CLINICAL TRIAL: NCT05066282
Title: Long-Term Safety and Persistence of Effectiveness of Manualized MDMA-Assisted Therapy for the Treatment of Posttraumatic Stress Disorder
Brief Title: Long-Term Safety and Effectiveness of MDMA-Assisted Therapy for PTSD
Acronym: MPLONG
Status: Completed | Type: Observational
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: MPLONG
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with past PTSD who received IMP in the main study: Non-interventional follow-up study

SUMMARY:
The goal of this long-term follow-up study is to measure how long effects of MDMA-assisted therapy last in participants with PTSD who were treated in a prior Phase 3 clinical trial of MDMA-assisted therapy.

The main question it aims to answer is: Does MDMA-assisted therapy result in lasting reductions in PTSD symptoms?

Participants who have received at least one dose of MDMA-assisted therapy will take a PTSD assessment at least six months after their last MDMA-assisted therapy session in the main study.

DETAILED DESCRIPTION:
This non-interventional study will serve as the long-term follow-up (LTFU) protocol for MDMA-assisted therapy clinical trials and will measure persistence of effectiveness using the CAPS-5 as a measure of PTSD symptom severity. The primary objective of this study is to evaluate the long-term effectiveness of MDMA-assisted therapy for treatment of PTSD as measured by the change in CAPS-5 Total Severity Score (actual or imputed) from the main study Baseline and Study Termination to LTFU IR Assessments (Visit 1). Additionally, this study will gather data to support health economics and cost effectiveness analyses of this treatment. Participants who have received at least one dose of Investigational Medicinal Product (IMP) in the main study will be eligible to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in a MAPS-sponsored study of MDMA-assisted therapy for the treatment of PTSD
2. Have received Investigational Medicinal Product (IMP) in at least one Experimental Session in the main study
3. Agree to be contacted by study team at least six months after the last Experimental Session in the main study to schedule and participate in LTFU visits

Exclusion Criteria:

1. Are not able to give adequate informed consent
2. Have any current problem which, in the opinion of the investigator or Medical Monitor, might interfere with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with past posttraumatic stress disorder (PTSD) who have completed at least one Experimental Session in the main study protocol.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-V (CAPS-5) Total Severity Score (actual or imputed) from the main study Baseline and Study Termination to assessment in the current LTFU study | LTFU IR Assessments at Least 6 Months Since Last Experimental Session in Main Study (Visit 1)
  The Clinician-Administered PTSD Scale for DSM-V (CAPS-5) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-5. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mitchell, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- USCF, San Francisco, California, United States
- Dr. Simon Amar Inc, Montreal, Quebec, Canada
- Israel (2):
  - Beer Yaakov Mental Health Center, Be’er Ya‘aqov
  - Tel Hashomer, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT05066282/ICF_000.pdf